CLINICAL TRIAL: NCT06788808
Title: The Role of Ultrasonography in Pregnancy in the Study of Fetal Central Nervous System Malformations
Acronym: CNS_2021
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CNS_2021
Record Dates: First submitted 2024-12-03; First posted 2025-01-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-10

CONDITIONS: Malformation Brain
Keywords: Prenatal ultrasounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fetus with CNS malformations: Evaluation of ultrasound images routinely performed during pregnancy in fetuses with brain malformation
  Interventions: Other: Comparison between groups
- Fetus withous CNS malformations: Evaluation of ultrasound images routinely performed during pregnancy in healthy fetuses
  Interventions: Other: Comparison between groups

INTERVENTIONS:
Other: Comparison between groups — Ultrasound images acquired during routine ultrasound scans performed in healthy fetuses and in fetuses found to have CNS malformations will be reviewed. Ultrasound images acquired from January 2000 to May 2021 will be analyzed until a sample size of approximately 80 patients is reached, who will be divided into 2 groups: group A (patients whose fetus has CNS malformations) and group B (healthy patients whose fetus has no anatomical CNS abnormalities).

SUMMARY:
The aim of this observational study is to evaluate the correlation between new ultrasound patterns and fetal central nervous system (CNS) malformations.

DETAILED DESCRIPTION:
During fetal life, the CNS undergoes major changes, so it is important to study the evolution of brain morphology serially during intrauterine life.

Despite numerous data in the literature, prenatal ultrasound diagnosis of CNS malformations is often difficult due to the presence of imaging pictures that are nondiagnostic or difficult to interpret. Moreover, only some of the sonographic features of CNS malformations have been described in detail. Therefore, it is essential to study and describe the ultrasound pictures in order to identify new ultrasound patterns useful to identify the fetal malformation more clearly. Therefore, this study aims to retrospectively analyze the ultrasound images of fetuses with established brain malformations and compare them with those of healthy fetuses in order to highlight the presence of new ultrasound patterns, which may more clearly define the malformative pathology.

Ultrasound images routinely performed in pregnancy in fetuses with brain malformation and in healthy fetuses will be reviewed.

For each patient, information will be collected on:

* Age
* Previous pregnancies and their outcome
* Pregnancy arising spontaneously or through Medically Assisted Procreation techniques
* Family history of congenital malformation
* Type of central nervous system malformation (neural tube defects, holoprosencephaly, corpus callosum agenesis, cerebellar malformations, posterior cranial fossa cysts, other malformations)
* Gestational age at the time of diagnostic suspicion
* Gestational epoch at the time of diagnosis
* Pregnancy outcome (miscarriage, voluntary termination of pregnancy, spontaneous delivery or cesarean section)
* Presence of associated abnormalities affecting other anatomical districts

For each newborn, information will be collected on:

* Sex
* Weight
* Umbilical artery pH
* APGAR index at 5 and 10 minutes
* Neurological assessment in the immediate postpartum period
* Perinatal mortality

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years with single pregnancy and fetus with ultrasound diagnosis of central nervous system malformation (group A)
* Women with single pregnancy and normoconformed fetuses (group B).

Exclusion Criteria:

* Twin pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be divided into 2 groups: group A (patients whose fetus has central nervous system malformations) and group B (healthy patients whose fetus has no anatomical abnormalities of the central nervous system).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between new ultrasound patterns and fetal CNS malformations | up to 100 weeks
  Retrospectively analyze ultrasound images of fetuses with established brain malformations

SECONDARY OUTCOMES:
Comparison of ultrasound patterns found in fetuses with and without CNS malformations | up to 100 weeks
  Comparison of ultrasound scans of fetuses with and without CNS malformation to discover of new ultrasound patterns, which may more clearly define the malformative pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Pilu, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy